CLINICAL TRIAL: NCT00604539
Title: Study of the Effect of Chondroitin Sulphate on Synovial Inflammation in Patients With Osteoarthritis of the Knee
Brief Title: Effect of Chondroitin Sulphate on Synovial Inflammation in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioiberica (Industry)
Responsible Party: Dr. Josep Vergés, Scientific Medical Director, Bioibérica S.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS/IV-SIN-01; CS/IV-SIN-01
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Synovitis; Osteoarthritis; Joint Diseases; Muskuloskeletal Diseases
Keywords: Chondroitin sulphate; Synovitis; Knee osteoarthritis; Magnetic Resonance Imaging
MeSH Terms: conditions — Synovitis; Osteoarthritis; Joint Diseases; Osteoarthritis, Knee | interventions — Chondroitin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Chondroitin sulphate
  Interventions: Drug: Chondroitin sulphate (Condrosan)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chondroitin sulphate (Condrosan) — 800 mg (two capsules of 400 mg each) taken once a day for one year
  Arms: 1
Drug: Placebo — Two placebo capsules taken once a day for six months followed by an additional six month treatment of 800 mg (two capsules of 400 mg of Chondroitin sulphate each) taken once a day
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of a chondroitin sulphate conventional treatment on the degree of severity of synovitis, as measured by magnetic resonance in patients with knee OA with clinical synovitis.

ELIGIBILITY:
Inclusion Criteria:

* Primary OA of the knee according to ACR with synovitis criteria (warmth, swelling or effusion);
* OA of radiological stages 2 and 3 according to Kellgren-Lawrence;
* Minimum joint space width ≥2 mm in the medial femorotibial compartment on standing knee X-ray;
* VAS of pain while walking ≥40 mm.

Exclusion Criteria:

* Known allergy to chondroitin sulphate;
* Progressive or serious pathologies (cancer, AIDS,...);
* Other bone and articular diseases (antecedents and/or current signs) such as chondrocalcinosis, Paget's disease, rheumatoid arthritis, aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, hemochromatosis, Wilson's disease, osteochondromatosis;
* Corticosteroids (oral, injectable), indomethacin, therapeutic dose of glucosamine or chondroitin sulphate during the 12 weeks preceding inclusion;
* Hyaluronic Acid (intra-articular pathway) during the 26 weeks preceding inclusion;
* Radioactive synovectomy during the 12 weeks preceding inclusion;
* If the patient is receiving NSAID at baseline (D0), it should be maintained at a stable dosage as much as possible from D0 to D180. In the open phase of the study (D180 to D360), NSAID will also be allowed as rescue medication along with acetaminophen.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the change in the severity of synovitis measured by MRI according to the modified methods of Loeuille et al. after chondroitin sulphate treatment in patients with knee OA and clinical signs of synovitis | One year

SECONDARY OUTCOMES:
Changes of cartilage volume and subchondral bone lesions | One year
Pain measured by VAS | One year
WOMAC index | One year
SF-36 Health Questionaire | One year
Assessment of joint swelling, effusion | One year
Use of rescue medication | One year
Tolerability | One year
Adverse events | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Pelletier, Prof., Dr., Principal Investigator — ArthroLab Inc.; Johanne Martel-Pelletier, Prof., Dr., Principal Investigator — ArthroLab Inc.
Locations (4):
- Canada (4):
  - Inst. De Rhumatologie, Montreal, Quebec
  - Groupe de recherche en rhumatologie et maladies osseuses, Ste-Foy, Quebec
  - Centre de rhumatologie St-Louis, Ste-Foy, Quebec
  - Centre de recherche musculo-squelettique, Trois-Rivières, Quebec

REFERENCES:
- [Background] Berthiaume MJ, Raynauld JP, Martel-Pelletier J, Labonte F, Beaudoin G, Bloch DA, Choquette D, Haraoui B, Altman RD, Hochberg M, Meyer JM, Cline GA, Pelletier JP. Meniscal tear and extrusion are strongly associated with progression of symptomatic knee osteoarthritis as assessed by quantitative magnetic resonance imaging. Ann Rheum Dis. 2005 Apr;64(4):556-63. doi: 10.1136/ard.2004.023796. Epub 2004 Sep 16. PMID 15374855
- [Background] Fajardo M, Di Cesare PE. Disease-modifying therapies for osteoarthritis : current status. Drugs Aging. 2005;22(2):141-61. doi: 10.2165/00002512-200522020-00005. PMID 15733021
- [Background] Clegg DO, Reda DJ, Harris CL, Klein MA, O'Dell JR, Hooper MM, Bradley JD, Bingham CO 3rd, Weisman MH, Jackson CG, Lane NE, Cush JJ, Moreland LW, Schumacher HR Jr, Oddis CV, Wolfe F, Molitor JA, Yocum DE, Schnitzer TJ, Furst DE, Sawitzke AD, Shi H, Brandt KD, Moskowitz RW, Williams HJ. Glucosamine, chondroitin sulfate, and the two in combination for painful knee osteoarthritis. N Engl J Med. 2006 Feb 23;354(8):795-808. doi: 10.1056/NEJMoa052771. PMID 16495392
- [Background] Hochberg MC, Altman RD, Brandt KD, Clark BM, Dieppe PA, Griffin MR, Moskowitz RW, Schnitzer TJ. Guidelines for the medical management of osteoarthritis. Part II. Osteoarthritis of the knee. American College of Rheumatology. Arthritis Rheum. 1995 Nov;38(11):1541-6. doi: 10.1002/art.1780381104. PMID 7488273
- [Background] Leeb BF, Schweitzer H, Montag K, Smolen JS. A metaanalysis of chondroitin sulfate in the treatment of osteoarthritis. J Rheumatol. 2000 Jan;27(1):205-11. PMID 10648040
- [Background] Loeuille D, Chary-Valckenaere I, Champigneulle J, Rat AC, Toussaint F, Pinzano-Watrin A, Goebel JC, Mainard D, Blum A, Pourel J, Netter P, Gillet P. Macroscopic and microscopic features of synovial membrane inflammation in the osteoarthritic knee: correlating magnetic resonance imaging findings with disease severity. Arthritis Rheum. 2005 Nov;52(11):3492-501. doi: 10.1002/art.21373. PMID 16255041
- [Background] McAlindon TE, LaValley MP, Gulin JP, Felson DT. Glucosamine and chondroitin for treatment of osteoarthritis: a systematic quality assessment and meta-analysis. JAMA. 2000 Mar 15;283(11):1469-75. doi: 10.1001/jama.283.11.1469. PMID 10732937
- [Background] Michel BA, Stucki G, Frey D, De Vathaire F, Vignon E, Bruehlmann P, Uebelhart D. Chondroitins 4 and 6 sulfate in osteoarthritis of the knee: a randomized, controlled trial. Arthritis Rheum. 2005 Mar;52(3):779-86. doi: 10.1002/art.20867. PMID 15751094
- [Background] Morreale P, Manopulo R, Galati M, Boccanera L, Saponati G, Bocchi L. Comparison of the antiinflammatory efficacy of chondroitin sulfate and diclofenac sodium in patients with knee osteoarthritis. J Rheumatol. 1996 Aug;23(8):1385-91. PMID 8856618
- [Background] Zhang W, Doherty M, Arden N, Bannwarth B, Bijlsma J, Gunther KP, Hauselmann HJ, Herrero-Beaumont G, Jordan K, Kaklamanis P, Leeb B, Lequesne M, Lohmander S, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Swoboda B, Varatojo R, Verbruggen G, Zimmermann-Gorska I, Dougados M; EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). EULAR evidence based recommendations for the management of hip osteoarthritis: report of a task force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2005 May;64(5):669-81. doi: 10.1136/ard.2004.028886. Epub 2004 Oct 7. PMID 15471891
- [Background] Raynauld JP, Martel-Pelletier J, Berthiaume MJ, Beaudoin G, Choquette D, Haraoui B, Tannenbaum H, Meyer JM, Beary JF, Cline GA, Pelletier JP. Long term evaluation of disease progression through the quantitative magnetic resonance imaging of symptomatic knee osteoarthritis patients: correlation with clinical symptoms and radiographic changes. Arthritis Res Ther. 2006;8(1):R21. doi: 10.1186/ar1875. Epub 2005 Dec 30. PMID 16507119
- [Background] Richy F, Bruyere O, Ethgen O, Cucherat M, Henrotin Y, Reginster JY. Structural and symptomatic efficacy of glucosamine and chondroitin in knee osteoarthritis: a comprehensive meta-analysis. Arch Intern Med. 2003 Jul 14;163(13):1514-22. doi: 10.1001/archinte.163.13.1514. PMID 12860572
- [Background] Uebelhart D, Malaise M, Marcolongo R, de Vathaire F, Piperno M, Mailleux E, Fioravanti A, Matoso L, Vignon E. Intermittent treatment of knee osteoarthritis with oral chondroitin sulfate: a one-year, randomized, double-blind, multicenter study versus placebo. Osteoarthritis Cartilage. 2004 Apr;12(4):269-76. doi: 10.1016/j.joca.2004.01.004. PMID 15023378
- [Result] Wildi LM, Raynauld JP, Martel-Pelletier J, Beaulieu A, Bessette L, Morin F, Abram F, Dorais M, Pelletier JP. Chondroitin sulphate reduces both cartilage volume loss and bone marrow lesions in knee osteoarthritis patients starting as early as 6 months after initiation of therapy: a randomised, double-blind, placebo-controlled pilot study using MRI. Ann Rheum Dis. 2011 Jun;70(6):982-9. doi: 10.1136/ard.2010.140848. Epub 2011 Mar 1. PMID 21367761